CLINICAL TRIAL: NCT02581475
Title: Efficacy of Segmental Examination Twice of Proximal Colon on Adenoma Detection: a Prospective, Randomized, Controlled Study
Brief Title: Efficacy of Segmental Examination Twice of the Proximal Colon on Adenoma Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yanqing Li (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, Professor, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2015SDU-QILU-G12
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-08

CONDITIONS: Colonic Polyps
Keywords: Adenoma detection rate; Colonoscopy; Withdrawal time
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Extending withdrawal time in the proximal colon: After cecal intubation, the colonoscopy is withdrawn to the hepatic flexure and then to the splenic flexure with an extended withdrawal time during colonoscopy.
  From cecum to hepatic flexure, 1.5-2 min is required and 2.5-3 min is required from heptic flexure to splenic flexure.
  Interventions: Procedure: Extending withdrawal time in the proximal colon
- Group B (Experimental): Segmental examination twice of the proximal colon: After cecal intubation, the colonoscopy is withdrawn to the hepatic flexure and then the colonoscopy is intubated to the cecum again. The same procedure is performed in the colonic segment from hepatic flexure to splenic flexure. The withdrawal time in each colonic segment is similar to the group A.
  Interventions: Procedure: Segmental examination twice of the proximal colon

INTERVENTIONS:
Procedure: Extending withdrawal time in the proximal colon
  Arms: Group A
Procedure: Segmental examination twice of the proximal colon
  Arms: Group B

SUMMARY:
Segmental examination twice of the proximal colon might be helpful to increase adenoma detection rate (ADR).

DETAILED DESCRIPTION:
Colonoscopy is the gold standard screening test for colorectal cancer (CRC). Removal of adenomas can reduce the incidence and mortality of CRC. However, there is evidence that some patients may develop interval cancers-cancers developed within 3-5 years following colonoscopy and polypectomy. The overall rate of interval cancer was 1.1-2.7 per 1000 person-years. Several studies have suggested that patients who develop interval cancers are more likely to have proximal compared than distal cancers.

One hypothesis is that adenomas may be more likely to be missed in the proximal colon compared with the distal colon. Serrated polyps and some adenomas in the proximal colon may be difficult to detect if they are flat, covered with mucus, or behind folds. A second hypothesis is that neoplastic lesions of the proximal colon may biologically differ from distal lesions and progress to malignancy with a short dwell time.

Several tandem back to back colonoscopy studies have demonstrated that up to 27% adenomas in the proximal colon are missed during routine screening colonoscopy. Hover, examining the colon twice as that in the back to back studies is difficult to be performed in clinical practice. Thus, we developed a novel colonoscopy technique, segmental examination twice of the proximal colon, that is simple and easy to be performed. The current study aims to examine the efficacy of segmental examination twice of the proximal colon on adenoma detection rate (ADR) during routine screening and surveillance colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Asia-Pacific Colorectal Screening score ≥2, such as patients ≥ 50 years, patients with a family history of colorectal cancer in a first-degree relative or male patients with current or past smoking.

Exclusion Criteria:

* Patients with prior resection of the proximal colon, advanced colonic cancer, inflammatory bowel disease, or polyposis syndrome.
* The cecum could not be intubated.
* Inadequate bowel preparation (Boston Bowel Preparation Scale score <2 in any segment of the colon).
* Biopsies were not available.
* Unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD, MD, Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong Province, China
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Martinez ME, Baron JA, Lieberman DA, Schatzkin A, Lanza E, Winawer SJ, Zauber AG, Jiang R, Ahnen DJ, Bond JH, Church TR, Robertson DJ, Smith-Warner SA, Jacobs ET, Alberts DS, Greenberg ER. A pooled analysis of advanced colorectal neoplasia diagnoses after colonoscopic polypectomy. Gastroenterology. 2009 Mar;136(3):832-41. doi: 10.1053/j.gastro.2008.12.007. Epub 2008 Dec 9. PMID 19171141
- [Background] Butterly L, Robinson CM, Anderson JC, Weiss JE, Goodrich M, Onega TL, Amos CI, Beach ML. Serrated and adenomatous polyp detection increases with longer withdrawal time: results from the New Hampshire Colonoscopy Registry. Am J Gastroenterol. 2014 Mar;109(3):417-26. doi: 10.1038/ajg.2013.442. Epub 2014 Jan 7. PMID 24394752
- [Background] Heresbach D, Barrioz T, Lapalus MG, Coumaros D, Bauret P, Potier P, Sautereau D, Boustiere C, Grimaud JC, Barthelemy C, See J, Serraj I, D'Halluin PN, Branger B, Ponchon T. Miss rate for colorectal neoplastic polyps: a prospective multicenter study of back-to-back video colonoscopies. Endoscopy. 2008 Apr;40(4):284-90. doi: 10.1055/s-2007-995618. PMID 18389446
- [Derived] Guo CG, Zhang F, Ji R, Li Y, Li L, Zuo XL, Li YQ. Efficacy of segmental re-examination of proximal colon for adenoma detection during colonoscopy: a randomized controlled trial. Endoscopy. 2017 Mar;49(3):243-250. doi: 10.1055/s-0042-122013. Epub 2017 Jan 27. PMID 28129661

RESULTS

PARTICIPANT FLOW:
Groups:
- Extending Withdrawal Time: After cecal intubation, the colonoscopy is withdrawn to the hepatic flexure and then to the splenic flexure with an extended withdrawal time during colonoscopy.
- Segmental Examination Twice: After cecal intubation, the colonoscopy is withdrawn to the hepatic flexure and then the colonoscopy is intubated to the cecum again. The same procedure is performed in the colonic segment from hepatic flexure to splenic flexure.
Period: Overall Study
Arm/Group | Extending Withdrawal Time | Segmental Examination Twice
Started | 193 | 193
Completed | 182 | 178
Not Completed | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extending Withdrawal Time | Segmental Examination Twice | Total
Number analyzed (Participants) | 182 | 178 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (10.3) | 55.0 (11.0) | 54.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 83 | 163
  Male | 102 | 95 | 197

OUTCOME MEASURES:

1. Primary Outcome: Difference of Adenoma Detection Rate in the Proximal Colon Among 2 Group.
Description: Adenoma detection rate in the proximal colon was the proportion of participants wiht more than one adenomas in proximal colon.
Time Frame: During routine screening and surveillance colonoscopy, for up to 1 hour, number of adenomas was recorded. About 1 month after this study, adenoma detetion rates were calculated.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Extending Withdrawal Time | Segmental Examination Twice
Number analyzed (Participants) | 182 | 178
proportion of participants | 0.236 [0.175 to 0.298] | 0.331 [0.262 to 0.4]

2. Secondary Outcome: Withdrawal Time in the Proximal Colon Among 2 Group.
Time Frame: During routine screening and surveillance colonoscopy, for up to 1 hour, withdrawal time was recorded. About 1 month after this study, mean withdrawal time was calculated.
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Extending Withdrawal Time | Segmental Examination Twice
Number analyzed (Participants) | 182 | 178
minute | 4.34 (1.36) | 4.29 (1.23)

3. Secondary Outcome: Duration of the Total Colonoscopy Among 2 Group.
Time Frame: During routine screening and surveillance colonoscopy, for up to 1 hour, the duration of colonoscopy was recorded. About 1 month after this study, mean duration of the colonoscopy was calculated.
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Extending Withdrawal Time | Segmental Examination Twice
Number analyzed (Participants) | 182 | 178
minute | 16.98 (4.92) | 17.45 (5.25)

4. Secondary Outcome: Adenomas Per Patient in the Proximal Colon Among 2 Group.
Time Frame: During routine screening and surveillance colonoscopy, for up toafter 1 hour, the number of adenomas was recorded. About 1 month after this study, mean number of adenomas in proximal colon was calculated.
Measure: Mean (Standard Deviation); unit: adenomas per patient
Arm/Group | Extending Withdrawal Time | Segmental Examination Twice
Number analyzed (Participants) | 182 | 178
adenomas per patient | 0.36 (0.704) | 0.54 (0.921)

ADVERSE EVENTS:
Arm/Group | Extending Withdrawal Time | Segmental Examination Twice
Serious Adverse Events (participants affected / at risk) | 0/182 | 0/178
Other Adverse Events (participants affected / at risk) | 0/182 | 0/178

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No